CLINICAL TRIAL: NCT00973297
Title: A Targeted Falls Prevention Program in Rehabilitation In-Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: YORAM MAARAVI MD, HADASSAH MEDICAL ORGANIZATION
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 151059-HMO-CTIL
Record Dates: First submitted 2009-08-25; First posted 2009-09-09 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: Accidental Falls
Keywords: Falls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Falls prevention (Experimental)
  Interventions: Other: Multidisciplinary falls prevention
- Control group (No Intervention): Routine rehabilitation treatment

INTERVENTIONS:
Other: Multidisciplinary falls prevention — Group education on falls risk and mobility and transfers safety; Physical therapy at the subjects' bedside consisting of balance training; Medical assessment - medications use (anxiolytics/hypnotics, neuroleptics, antihypertensives, antiarrhythmics and other vasodilators) with effort to discontinue or reduce dose when possible; orthostatic hypotension - discontinue/reduce dose of related medications; urinary frequency/incontinence - evaluation and treatment; delirium - evaluation and treatment; visual pathology - evaluation and treatment
  Arms: Falls prevention

SUMMARY:
Falls are a major complication in patients treated in rehabilitation departments, yet studies evaluating different interventions to reduce falls-risk are rare and inconclusive.

The aim of the present study is to evaluate the efficacy of a multidisciplinary fall-prevention program to reduce falls and injury in stroke patients treated in a rehabilitation department.

All stroke patients consecutively admitted to the department of rehabilitation at Hadassah-Hebrew University Medical Center for a period of one year will be eligible for inclusion. Upon receiving an informed consent subjects will be randomized to the intervention group or the control (convention care) group.

There are no exclusion criteria. The Intervention includes group education on risk of falling and safe mobility and transfers; physical therapy of balance training at the patients' bedside twice weekly and medical assessment of medication use (anxiolytics/hypnotics, neuroleptics, antihypertensives and other vasodilators), orthostatic hypotension, urinary frequency/incontinence, delirium and visual problems.

Intervention therapy will not be given as an extra time, rather at the same treatment time as the control group.

Primary outcomes are rate of falls and related injuries.

ELIGIBILITY:
Inclusion Criteria:

* All stroke patients admitted to rehabilitation

Exclusion Criteria:

* None

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-11 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Rate of falls and fall-related injury | At one year

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Maaravi, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel